CLINICAL TRIAL: NCT07145333
Title: Explore the Relationship Between Single Nucleotide Polymorphisms and Topotecan Response and Toxicity in Patients With Small Cell Lung Cancer.
Brief Title: Pharmacogenomics ANDA SNP Clinical Study - Topotecan and Single Nucleotide Polymorphisms
Acronym: Drug-SNP
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Collaborators: UnitedHealthcare (Other)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IORG Director, Medical Monitor, Safety Officer, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IND 178174 Commercial; FWA00015357 (Registry Identifier: HHS, Human Protections Administrator); NPI-1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI-1023387701 (Registry Identifier: HHS, Health Care Provider Organization); IRB00009424 (Registry Identifier: HHS, IRB); IORG0007849 (Registry Identifier: HHS, IORG); IND178174 (Registry Identifier: FDA, IND)
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: SCLC
Keywords: SNP; Topotecan; TOPO; CYP; Genotype
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: * The usual approach group (Oral)
  * The study approach group (Oral) (China Import)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No-placebo and random and double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topotecan - usual (Experimental): * Topotecan Capsule
  * Chemotherapy
  * Topotecan Capsule
  * Usual Approach Group
  Interventions: Drug: Topotecan - usual
- Topotecan - study (Experimental): * China Import Topotecan Capsule
  * Chemotherapy
  * China Import Topotecan Capsule
  * Study Approach Group
  Interventions: Drug: Topotecan - study

INTERVENTIONS:
Drug: Topotecan - usual — Topotecan Capsule
  Other Names: Usual Topotecan Capsule Chemotherapy
  Arms: Topotecan - usual
Drug: Topotecan - study — China Import Topotecan Capsule
  Other Names: Study Topotecan Capsule Chemotherapy
  Arms: Topotecan - study

SUMMARY:
Explore the relationship between drug target topoisomerase I gene single nucleotide polymorphisms and Topotecan therapeutic-effects in patients with small cell lung cancer, based on Oxford precisely sequencing drug targets' genes.

Explore the relationship between drug target CYP4503A4 gene single nucleotide polymorphisms and Topotecan side-effects in patients with small cell lung cancer, based on Oxford precisely sequencing drug targets' genes.

DETAILED DESCRIPTION:
The usual approach group, after lung tissue biopsy, 300 double blind random group separated SCLC patients currently used the Chemotherapy on Topotecan capsule, it will try to look for the relationship between the Topotecan therapeutic efficacy and the Topoisomerase I SNP Genotyping, and the relationship between the Topotecan therapeutic safety and the CYP4503A4 SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

The study approach group, after lung tissue biopsy, 300 double blind random group separated SCLC patients currently used the Chemotherapy on China Import Topotecan Capsule, it will try to look for the relationship between the Topotecan therapeutic efficacy and the Topoisomerase I SNP Genotyping, and the relationship between the Topotecan therapeutic safety and the CYP4503A4 SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

1. Detect drug target whole gene precision sequence of everyone patient for all 600 recruited double blind SCLC patients.
2. Mutually compare everyone patient drug target whole gene precision sequence for a total of 600 recruited double blind SCLC patients.
3. Calculate drug target gene SNPs in all 600 recruited double blind SCLC patients.
4. Correlate everyone patient drug target gene SNP to everyone patient drug efficacy.
5. Correlate everyone patient drug target gene SNP to everyone patient drug safety.
6. Mutually compare the usual approach group SNPs (300 double blind random group separated SCLC patients) with the study approach group SNPs (300 double blind random group separated SCLC patients).
7. Confirm the relationship between drug target gene SNPs and drug efficacy.
8. Confirm the relationship between drug target gene SNPs and drug safety.

ELIGIBILITY:
* Select 600 Small Cell Lung Cancer Patients who are suitable for lung tissue biopsy
* Dosage Duration at least 45 days
* The usual approach group - Recruit 300 double blind random group separated SCLC patients currently used the Chemotherapy on Topotecan Capsule after lung tissue biopsy, like as the usual approach group.
* The study approach group - Recruit 300 double blind random group separated SCLC patients currently used the Chemotherapy on China Import Topotecan Capsule after lung tissue biopsy, like as the study approach group.

Inclusion Criteria:

* 1. Clinical diagnosis of Small Cell Lung Cancer (SCLC)
* 2. Clinical lung tissue biopsy diagnosis of SCLC
* 3. Suitable for enough lung tissue biopsy of SCLC
* 4. Random and double blind
* 5. Measurable disease
* 6. Adequate organ functions
* 7. Adequate performance status
* 8. Age 24 years old and over
* 9. Sign an informed consent form
* 10. Receive blood-drawing

Exclusion Criteria:

* 1. Pneumonectomy
* 2. Treatment with other anti-cancer therapies and cannot be stopped currently
* 3. Pregnancy
* 4. Breast-feeding
* 5. The patients with other serious intercurrent illness or infectious diseases
* 6. Have more than one different kind of cancer at the same time
* 7. Serious Allergy to Drugs
* 8. Clot or Bleed Tendency
* 9. Serious Risks or Serious Adverse Events of the drug product
* 10. The prohibition of drug products
* 11. Have no therapeutic effects
* 12. Follow up to the most current label

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Find Topotecan Drug Targets' SNP Genotypes which are effectiveness-associated, and which are risk-associated. | Duration up to 14 weeks
  1. Recruit 300 double blind random group separated SCLC patients currently used the Chemotherapy on Topotecan Capsule after lung tissue biopsy, like as the usual approach group.
  2. Recruit 300 double blind random group separated SCLC patients currently used the Chemotherapy on China Import Topotecan Capsule after lung tissue biopsy, like as the study approach group.
  3. Assay above every SCLC patient-specific Topotecan drug target (Topoisomerase I) SNP genotype in his or her WBC cell whole genome DNA with Oxford precisely sequencing.
  4. Assay above every SCLC patient-specific Topotecan drug target (CYP4503A4) SNP genotype in his or her WBC cell whole genome DNA with Oxford precisely sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: HAN XU, MD/PhD/FAPCR, Study Chair — Medicine Invention Design, Inc. - IRB00009424 - IORG0007849; HAN XU, MD/PhD/FAPCR, Study Director — Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701; HAN ID XU, MD/PhD/FAPCR, Principal Investigator — Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701
Locations (1):
- Medicine Invention Design Incorporation, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FWA < 00015357 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search
- See also: IRB < 00009424 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search
- See also: IORG < 0007849 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search

DOCUMENTS (3):
  • Study Protocol (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT07145333/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT07145333/SAP_001.pdf
  • Informed Consent Form (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT07145333/ICF_002.pdf